CLINICAL TRIAL: NCT00471848
Title: Prospective Phase II Study of Rabbit Antithymocyte Globulin (ATG, Thymoglobuline®, Genzyme) With Ciclosporin for Patients With Acquired Aplastic Anaemia and Comparison With Matched Historical Patients Treated With Horse ATG and Ciclosporin
Brief Title: Rabbit Antithymocyte Globulin (Thymoglobuline) With Ciclosporin for Patients With Acquired Aplastic Anaemia
Acronym: RATGAA07
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2007-000902-55; RATGAA07
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Results first posted 2021-10-18 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Aplastic Anemia
Keywords: Thymoglobuline; Rabbit ATG; Ciclosporin; Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Antithymocyte globulin with cyclosporin in first line treatment of patients with acquired severe aplastic anaemia and patients with non-severe aplastic anaemia who are transfusion dependent
  Interventions: Drug: rabbit antithymocyte globulin

INTERVENTIONS:
Drug: rabbit antithymocyte globulin — 1.5 vials/10kg daily for 5 days
  Other Names: Thymoglobuline

SUMMARY:
To assess the tolerability and effectiveness of rabbit antithymocyte globulin (ATG, Thymoglobuline) with ciclosporin in the first line treatment of patients with acquired severe aplastic anaemia, and patients with non-severe aplastic anaemia and who are transfusion dependent.

DETAILED DESCRIPTION:
Traditionally horse antithymocyte globulin (ATG) has been the preferred animal source of ATG as first line treatment for acquired aplastic anaemia (AA) patients who are ineligible for bone marrow transplantation (BMT). For severe AA (SAA) the combination of ATG and Ciclosporin (CSA) results in response in 60-75% of patients and the response is superior to using either agent alone. The addition of granulocyte colony stimulating factor (G-CSF) to the combination of ATG and CSA has so far shown no significant benefit in terms of response and survival, but an European Group for Blood and Marrow Transplantation (EBMT) prospective study is currently evaluating this further in a larger number of patients. For patients with non-severe aplastic anaemia (NSAA) who are transfusion dependent, the combination of ATG and CSA was shown to be superior to CSA alone in an EBMT prospective randomised study, with a higher response rate, superior blood counts and improved disease free survival using the combination of ATG with CSA.

There have been no phase II studies of rabbit ATG (Thymoglobuline®) in the treatment of AA as first line therapy. Preliminary results from a small single centre study compared horse ATG (ATGAM) with rabbit ATG (Fresenius) in children and showed response rates of 93% and 47%, respectively, but it is likely that different preparations of rabbit ATG will vary in their efficacy. Rabbit ATG is more commonly used for a second course following relapse or lack of response to a first course of horse ATG. Rabbit ATG in combination with CSA and G-CSF was used in patients with SAA who had failed to respond to a course of horse ATG with CSA and G-CSF. Overall response (transfusion independence) was seen in 23/30 (77%) of patients after a median of 95 days and complete response (neutrophils > 2.0, haemoglobin > 11, and platelets > 100) in 9/30 (30%). Rabbit ATG was well tolerated; no anaphylaxis or severe side effects were reported. Another study of 43 patients treated with rabbit ATG and CSA following non-response or relapse after horse ATG and CSA, showed 30% response rate among non-responding patients and 65% response rate for relapsing patients.

Studies comparing the antibody specificities between Thymoglobuline® and Lymphoglobuline® are in broad agreement, but (a) Lymphoglobuline® has fewer studies and those reported are older, because the product is older and has been less extensively developed (b) antibodies against certain epitopes are inconsistently present (c) not all antibody specificities have been examined in some studies and (d) different methods of testing have been used. There is a view that it is the immunogen and not the animal species which is most important in creating differences between different ATGs.

ELIGIBILITY:
Inclusion Criteria:

1. Must fulfil definition of aplastic anaemia:

   There must be at least two of the following:
   * haemoglobin < 10g/dl
   * platelet count < 50 x 109/l
   * neutrophil count < 1.5 x 109/l, and a hypocellular bone marrow on bone marrow biopsy

   SAA as defined by a hypocellular bone marrow of <25% cellularity and two of the following:
   * neutrophil count < 0.5 x 109/l
   * platelets < 20 x 109/l
   * reticulocytes < 20 x 109/l

   NSAA as defined by a hypocellular bone marrow and cytopenia in at least two cell lines and neutrophil count > 0.5 x 109/l, and red cell and/or platelet transfusion dependence
2. Have acquired aplastic anaemia
3. Time from diagnosis to study registration maximum 6 months
4. No prior treatment except for haemopoietic growth factors given for no more than four weeks, and androgens
5. Age minimum 16 years with no upper age limit

Exclusion Criteria:

1. Eligibility for an human leukocyte antigens (HLA)-matched sibling donor transplant for SAA patients
2. Prior therapy with ATG or CSA
3. Haematopoeitic growth factors more than 4 weeks before study enrolment
4. Diagnosis of Fanconi anaemia, dyskeratosis congenita or congenital bone marrow failure syndrome
5. Evidence of myelodysplastic disease
6. Paroxysmal nocturnal haemoglobinuria with evidence of significant haemolysis, history of Paroxysmal Nocturnal Hemoglobinuria (PNH) associated thrombosis or a PNH clone >50% by flow cytometry
7. Diagnosis or previous history of carcinoma (except local cervical, basal cell, squamous cells, or melanoma)
8. Subject is pregnant (e.g. positive Human Chorionic Gonadotropin (HCG) test) or is breast feeding
9. Severe uncontrolled infection or unexplained fever >38 degrees Celsius
10. Subjects who have hepatic, renal cardiac, metabolic or other concurrent diseases of such severity that life expectancy is less than 3 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2011-10 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Marsh, Prof. MD., Principal Investigator — King's College Hospital NHS Trust
Locations (14):
- France (2):
  - Henri Mondor Hospital, Créteil
  - Hopital St. Louis, Paris
- Germany (4):
  - University Hospital Essen, Essen
  - University Hospital Eppendorf, Hamburg
  - Medical University Hannover, Hanover
  - Universitätsklinikum - Institut für klinische Transfusionsmedizin, Ulm
- Ospedale San Martino, Genova, Italy
- King Faisal Specialist Hospital & Research Cnetre, Riyadh, Saudi Arabia
- University Hospital, Basel, Switzerland
- United Kingdom (5):
  - Royal Bournemouth, Bournemouth
  - Addenbrooke's Hospital, Cambridge
  - St George's Hospital/ St George's University of London, London
  - King's College Hospital, London
  - Nottingham Universitry Hospital Trust, Nottingham

REFERENCES:
- [Result] Marsh JC, Bacigalupo A, Schrezenmeier H, Tichelli A, Risitano AM, Passweg JR, Killick SB, Warren AJ, Foukaneli T, Aljurf M, Al-Zahrani HA, Hochsmann B, Schafhausen P, Roth A, Franzke A, Brummendorf TH, Dufour C, Oneto R, Sedgwick P, Barrois A, Kordasti S, Elebute MO, Mufti GJ, Socie G; European Blood and Marrow Transplant Group Severe Aplastic Anaemia Working Party. Prospective study of rabbit antithymocyte globulin and cyclosporine for aplastic anemia from the EBMT Severe Aplastic Anaemia Working Party. Blood. 2012 Jun 7;119(23):5391-6. doi: 10.1182/blood-2012-02-407684. Epub 2012 Apr 27. PMID 22544699
- See also: Sponsor's website — http://www.ebmt.org
- See also: Publication — https://pubmed.ncbi.nlm.nih.gov/22544699/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 sites in 6 countries were open to include patients; in the end 10 sites entered all 35 patients. First Patient In (FPI) 04-Aug-2008, Last Patient In (LPI) 30-Sep-2010
Pre-assignment Details: Naive aplastic anaemia patients
Groups:
- Treatment Arm: Antithymocyte globulin with cyclosporin in first line treatment of patients with acquired severe aplastic anaemia and patients with non-severe aplastic anaemia who are transfusion dependent; the results were compared with historical controls from the European Group for Blood and Marrow Transplantation (EBMT) database. Patients were matched for age and disease status (NSAA, SAA, VSAA)
Period: Overall Study
Arm/Group | Treatment Arm
Started | 35
Completed | 35 (35 registered patients received the full 5-day Rabbit Antithymocyte Globulin (RATG) treatment)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Antithymocyte globulin with cyclosporin in first line treatment of patients with acquired severe aplastic anaemia and patients with non-severe aplastic anaemia who are transfusion dependent; the results were compared with historical controls from the EBMT database. Patients were matched for age and disease status (NSAA, SAA, VSAA)
Arm/Group | Treatment Arm
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 30
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response to Rabbit Antithymocyte Globulin (Thymoglobuline)
Description: Complete Response (CR) defined as:
  Haemoglobin normal for age and gender, neutrophils > 1.5 x 10E9/l, platelets > 150 x 10E9/l.
  Partial Response (PR) defined as:
  * transfusion independence (if previously dependent) or
  * doubling or normalisation of at least one cell line or
  * increase of baseline haemoglobin of > 3 g/dl (if initially <6) + neutrophils of > 0.5 x 10E9/l + platelets of > 20 x 10E9/l (if initially < 20)
  No Response (MR) is defined as: worse or not meeting criteria above
Time Frame: at 6months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 35
Participants
  CR | 1
  PR | 11
  NR | 18
  Transplanted | 3
  Dead | 2

2. Secondary Outcome: Failure Free and Overall Survival of Participants to Rabbit Antithymocyte Globulin (Thymoglobuline)
Description: Failure free survival is defined as a failure of the protocol: no achievement of response, relapse, disease progression requiring a second course of immune suppressive therapy (IST) or a stem cell transplant, death, or later clonal disorders such as Paroxysmal Nocturnal Hemoglobinuria (PNH), Myelodysplastic Syndrome (MDS) and Acute Myeloblastic Leukemia (AML).
Time Frame: at 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Experimental: Treament Arm: Antithymocyte globulin with cyclosporin in first line treatment of patients with acquired severe aplastic anaemia and patients with non-severe aplastic anaemia who are transfusion dependent
Arm/Group | Experimental: Treament Arm
Serious Adverse Events (participants affected / at risk) | 27/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Treament Arm (N=35)
Pyrexia (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Allergic Reaction / Hypersensitivy (Immune system disorders) | 1 (1)
Bacterial Infections (Infections and infestations) | 1 (1)
Bilateral Basal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood-reactivation (Infections and infestations) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Coccy geal fistula abscessed (Infections and infestations) | 1 (1)
Colonisation in Staphylococcus aures methicillin resistant (Infections and infestations) | 1 (1)
Death (General disorders) | 6 (6)
Disease progression (General disorders) | 2 (2)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Facial Infection (Infections and infestations) | 1 (1)
Elevated ALT levels (Investigations) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 5 (6)
Hyper Bilirubinimia (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Klebsiella Septicaemia (Infections and infestations) | 1 (1)
Hickmann Line Infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 5 (5)
Neutropenic Fever (Infections and infestations) | 1 (1)
Norovirus infection (Infections and infestations) | 1 (1)
Pyrexia with rigours (General disorders) | 1 (1)
Pancreatic endocrine, glucose intolerance (Endocrine disorders) | 1 (1)
Renal Impairment (Metabolism and nutrition disorders) | 1 (1)
Retinopathy (Eye disorders) | 1 (1)
Seizures (Nervous system disorders) | 1 (1)
Secondary Clonal Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sepsis (Infections and infestations) | 3 (4)
Serum Sickness (Immune system disorders) | 2 (2)
Unrelated Donor Stem Cell Transplant (General disorders) | 1 (1)
Vasovagal Episode (Cardiac disorders) | 1 (1)
Cholestasis (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participating PIs can not publish on the patients they have included in this prospective trial before the results of the trial have been published in a peer-reviewed journal.